CLINICAL TRIAL: NCT03893344
Title: Detection of STAT4 in Multiple Sclerotic Patients by Polymerase Chain Reaction and Flow Cytometry
Brief Title: STAT4 in Multiple Sclerosis by PCR and Flow Cytometry
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Mohammed SalahElDin, Assistant Lecturer at Assiut University, Assiut University
Other Study IDs: STAT4 gene in MS.
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: patients with Multiple Sclerosis in different stages diagnosed clinically according to revised McDonald's criteria 2010
  Interventions: Diagnostic Test: detection of STAT4 gene
- Control: Healthy peaple
  Interventions: Diagnostic Test: detection of STAT4 gene

INTERVENTIONS:
Diagnostic Test: detection of STAT4 gene — Individuals within both groups will be subjected to STAT4 gene polymorphism typing using both PCR and flow cytometry from a peripheral blood sample

SUMMARY:
1. To determine the level of STAT4 expression in different cases of multiple sclerosis and its relation to disease severity .
2. compare the sensitivity and specificity of STAT4 levels using both PCR and flow cytometry.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating and neurodegenerative disease of the central nervous system (CNS) (Huang et al., 2017).

The exact etiology of the disease is unknown, it is a heterogeneous, multifactorial and immune-mediated disease that is caused by complex gene-environment interactions (Olsson el al., 2017). It is mediated by autoreactive lymphocytes that cross the blood brain barrier (BBB) and enter the CNS where they cause local inflammation that results in demyelination, gliotic scarring, and axonal loss (Huang et al., 2017).

The onset of MS has been typically observed in individuals aged from 20 to 40 years, with the female to male ratio of 2:1 (Koch-Henriksen and Sørensen, 2010). According to a documented MS registry from Egypt done in 2010 and 2017, the epidemiology of MS was slightly differed from other Arab countries and western countries. The mean age of disease onset was 26.6±7.8 years, with the majority being females (2.11:1). Relapsing-remitting MS was the most common type (75.1%) (Hamdy et al., 2017). And its prevalence was found to be 14.1/100.000 (Hashem et al., 2010).

The pathological hallmark of MS is the accumulation of inflammatory demyelinating lesions that occur in the white matter and the grey matter of the brain and spinal cord (Celius and Smestad, 2009).

MS is regarded as a T cell mediated autoim¬mune disorder with a predominance of CD8+ cells compared with other T-cell subsets. The disease begins in inflammatory induced lesions consisting mainly of CD8+ T cells, and CD4+ T cells, and activate microglia/macrophages (Traugott et al., 1983; Ferguson el al., 1997). B lymphocytes and their cytokines are other factors in the pathogenesis of the disease. They have both positive and negative effects in the development of MS through lymphotoxin and IL-10, respectively (Duddy el al., 2007). It can be triggered by various environmental components, such as exposure to ultraviolet light, drugs, chemicals, and viral infections (Olsson el al., 2017).

The clinical symptoms of MS are determined by the exact neuroanatomical location of the plaque; the disease being essentially diagnosed by the manifestation of symptoms and signs attributable to lesions of white matter. It may appear as an abrupt onset of focal sensory disturbances that is accompanied by unilateral painless damage of vision, double vision, limb weakness, unsteadiness of gait, and bowel or bladder symptoms (Celius and Smestad, 2009).

Although MS is associated with change in average life expectancy, it is not considered a fatal condition and clinical course, which appears highly variable, is unpredictable for the individual patient. Typically, the early stages of disease ( relapsing remitting MS) (RRMS) are characterized by reversible clinical exacerbations, or relapses. It is caused by autoreactive immune cells that traffic into the CNS, resulting in focal inflammation and demyelination often visible as gadolinium-enhancing lesions on magnetic resonance imaging (MRI). Relapses are followed by periods of clinical remission as inflammation resolves and remyelination occurs (Mahad el al., 2015).

Secondary progressive MS (SPMS) is a chronic inflammation with scar formation, accumulation of axonal damage and brain atrophy, and inhibition of remyelination contribute to progressively worsening disability. In ~15% of patients, the disease is progressive from clinical onset and is designated as primary progressive MS (PPMS) (Harris et al., 2017).

The diagnosis of MS is primary clinical, to distinguish it from other similar neurological manifestations, McDonald criteria have been proposed (Filippi et al., 2018).

Intriguingly, genetically determined changes in signaling responses and activation thresholds in specific immune cell lineages have been described in MS. Identifying dysregulated signaling pathways in cell compartments relevant to the disease and their relationship with genetic variance could represent a useful strategy to better understand the natural history of MS and discover new therapeutic targets (Housley et el., 2015).

The human STAT (signal transducer and activator of transcription) genes have been identified in three chromosomal clusters: STAT1 and STAT4 on human chromosome 2 (q12-33); STAT2 and STAT6 on chromosome 12 (q13-14); and STAT3, STAT5a, and 5b on chromosome 17 (q11.2-22). This gene encodes a transcription factor that can be activated by interleukin (IL)-12 and IL-23 and plays a role in the signaling via type-1 interferon (IFN I) receptor (Ceccarelli et al., 2015).

STAT4 is essential for IL-12 signaling and induces interferon-gamma (IFNγ) production (Gestermann et al., 2010). Signal transmission from the interferons involves STAT1 and STAT4 (Raafat et al., 2015).

Abnormal levels of phosphorylated proteins belonging to the STAT family in the peripheral blood mononuclear cells of MS patients have been associated with a number of clinically relevant phenotypes (Canto et al., 2018).

The extensive involvement of type I and type II interferons in the pathogenesis of MS made STAT4 an obvious candidate region for genetic predisposition to these autoimmune diseases (Bolin et al. 2013). Moreover, the requirement of STAT4 in IL-23 induced IL-17 production has been suggested (Tanasescu et al. 2010).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of MS patients will be established clinically from the history according to revised McDonald's criteria 2010.

Exclusion Criteria:

* Patients proved not to have MS either at first interview or at any time during follow up or with other autoimmune diseases will be ruled out of the study.
* Healthy group with past or present medical history of autoimmune disease or other neurologic condition.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MS patients, fulfilling the inclusion criteria for the research, will be selected from Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
To determine the level of STAT4 expression in different cases of multiple sclerosis | baseline
  measuring the level of STAT4 gene in both the control group and different cases of multiple sclerotic and its relation to disease pathogenesis and severity

SECONDARY OUTCOMES:
compare the sensitivity and specificity of STAT4 levels using both PCR and flow cytometry. | baseline
  compare the sensitivity and specificity of STAT4 levels using both PCR and flow cytometry in peripheral blood sample which is easy and safe diagnostic method.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K Mostafa, Professor, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Housley WJ, Fernandez SD, Vera K, Murikinati SR, Grutzendler J, Cuerdon N, Glick L, De Jager PL, Mitrovic M, Cotsapas C, Hafler DA. Genetic variants associated with autoimmunity drive NFkappaB signaling and responses to inflammatory stimuli. Sci Transl Med. 2015 Jun 10;7(291):291ra93. doi: 10.1126/scitranslmed.aaa9223. PMID 26062845
- [Background] Filippi M, Bar-Or A, Piehl F, Preziosa P, Solari A, Vukusic S, Rocca MA. Multiple sclerosis. Nat Rev Dis Primers. 2018 Nov 8;4(1):43. doi: 10.1038/s41572-018-0041-4. PMID 30410033
- See also: Aberrant STAT phosphorylation signaling in peripheral blood mononuclear cells from multiple sclerosis patients. Journal of Neuroinflammation 15:72 — https://doi.org/10.1186/s12974-018-1105-9
- See also: Association of STAT4 polymorphism with severe renal insufficiency in lupus nephritis. PLoS One.8(12):e84450 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3873995/